CLINICAL TRIAL: NCT00681109
Title: Safety and Efficacy of Topical Interleukin-1-Receptor Antagonist in the Treatment of Signs and Symptoms of Posterior Blepharitis
Brief Title: Topical IL-1-Ra for Treatment of Posterior Blepharitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Reza Dana, MD (Other)
Responsible Party: Sponsor-Investigator, Reza Dana, MD, Principal Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-07-047
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Results first posted 2012-11-27 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Posterior Blepharitis
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Interleukin 1 Receptor Antagonist Protein; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Arm 1 (Active Comparator): 2.5% IL-1Ra
  Interventions: Drug: 2.5% IL-1Ra
- Placebo (Placebo Comparator): Artificial Tear
  Interventions: Drug: Placebo
- Treatment Arm 2 (Active Comparator): 5% IL-1Ra
  Interventions: Drug: 5% IL-1Ra

INTERVENTIONS:
Drug: 2.5% IL-1Ra — 2.5% custom made topical IL-1Ra three times a day in both eyes for three months
  Other Names: Anakinra 2.5%; Kineret 2.5%
  Arms: Treatment Arm 1
Drug: Placebo — custom eye drop to be applied three times a day in both eyes for three months
  Other Names: Artificial Tear
  Arms: Placebo
Drug: 5% IL-1Ra — 5% custom made topical IL-1Ra to both eyes 3 times a day for 3 months
  Other Names: Anakinra 5%; Kineret 5%
  Arms: Treatment Arm 2

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of Topical Interleukin-1-Receptor Antagonist in treatment of signs and symptoms of posterior blepharitis.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of posterior blepharitis
* A negative urine pregnancy test result for women of childbearing potential
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation
* Normal lid position and closure
* Ability to understand and provide informed consent to participate in this study
* Willingness to follow study instructions and likely to complete all required visits.

Exclusion Criteria:

* History of Stevens-Johnson syndrome or ocular pemphigoid
* History of eyelid surgery
* Intra-ocular surgery or ocular laser surgery within 3 months
* History of microbial keratitis, including herpes
* Active ocular allergies
* Corneal epithelial defect > 1mm2
* Use of topical steroids or Restasis within the past 2 weeks
* Use of tetracycline compounds (tetracycline, doxycycline, and minocycline) within the last month
* Use of isotretinoin (Accutane) within the past 6 months
* Have had any previous treatment with Anakinra (Kineret®) or any therapeutic agent targeted at IL-1 blockade
* Pregnant or lactating women
* Signs of current infection, including fever and current treatment with antibiotics
* Liver, renal, or hematologic disease
* The use of any other investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Dana, MD, MPH, MSc, Principal Investigator — Massachusetts Eye and Ear Infirmary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amparo F, Dastjerdi MH, Okanobo A, Ferrari G, Smaga L, Hamrah P, Jurkunas U, Schaumberg DA, Dana R. Topical interleukin 1 receptor antagonist for treatment of dry eye disease: a randomized clinical trial. JAMA Ophthalmol. 2013 Jun;131(6):715-723. doi: 10.1001/jamaophthalmol.2013.195. PMID 23599118

RESULTS

PARTICIPANT FLOW:
Groups:
- 2.5% IL-1Ra: Anakinra (IL-1Ra) 2.5% Topical Ophthalmic Solution three times per day.
- Placebo: Artificial Tear Topical Ophthalmic Solution three times per day.
- 5% IL-1Ra: Anakinra (IL-1Ra) 5% Topical Ophthalmic Solution three times per day.
Period: Overall Study
Arm/Group | 2.5% IL-1Ra | Placebo | 5% IL-1Ra
Started | 30 | 30 | 15
Completed | 28 | 24 | 15
Not Completed | 2 | 6 | 0
Not completed — Lost to Follow-up | 2 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2.5% IL-1Ra: Anakinra 2.5% Topical Ophthalmic Solution
- Placebo: Artificial Tear Topical Ophthalmic Solution
- 5% IL-1Ra: Anakinra 5% Topical Ophthalmic Solution
- Total: Total of all reporting groups
Arm/Group | 2.5% IL-1Ra | Placebo | 5% IL-1Ra | Total
Number analyzed (Participants) | 30 | 30 | 15 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14) | 53 (12) | 58 (16) | 52 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 10 | 44
  Male | 12 | 14 | 5 | 31
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 15 | 75
Meibomian Gland Secretion Quality [Mean (Standard Deviation); unit: units on a scale] — Meibomian Gland Secretion Quality has a range of 0 (normal secretion quality) to 3 (abnormal secretion quality)
  units on a scale | 1.9 (0.4) | 1.8 (0.5) | 1.9 (0.5) | 1.9 (0.5)
Tear Film Break-Up Time (TBUT) [Mean (Standard Deviation); unit: Seconds] — TBUT measures the amount of time, in seconds, that the tear film completely coats the ocular surface after each blink. The longer the time the tear film completely coats the ocular surface is considered to be better than a shorter amount of time.
  Seconds | 3.8 (2.8) | 3.8 (2.1) | 3.5 (2.2) | 3.7 (2.5)
Corneal Fluorescein Staining Score [Mean (Standard Deviation); unit: units on a scale] — CFS is used to assess the level of corneal epitheliopathy that is related to dry eye disease. The CFS scale ranges from 0 to 15 scale, with 0 representing the minimum level of corneal epitheliopathy and 15 representing the maximum level of epitheliopathy.
  units on a scale | 1.6 (0.9) | 1.7 (1.2) | 1.7 (0.9) | 1.7 (1.0)
Ocular Surface Disease Index (OSDI) [Mean (Standard Deviation); unit: units on a scale] — The Ocular Surface Disease Index (OSDI) is a 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning. OSDI is scored on a scale of 0 to 100, with higher scores representing greater disability.
  units on a scale | 44.2 (20.4) | 45.6 (21.1) | 48.5 (21.0) | 46.1 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: Meibomian Gland Secretion Quality
Description: Meibomian Gland Secretion Quality has a range of 0 (normal secretion quality) to 3 (abnormal secretion quality)
Time Frame: 12 Week Time Point
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 2.5% IL-1Ra | Placebo | 5% IL-1Ra
Number analyzed (Participants) | 30 | 30 | 15
Units on a scale | 1.7 (0.7) | 1.7 (0.4) | 1.8 (0.6)

2. Primary Outcome: Tear Breakup Time (TBUT)
Description: TBUT measures the amount of time, in seconds, that the tear film completely coats the ocular surface after each blink. The longer the time the tear film completely coats the ocular surface is considered to be better than a shorter amount of time.
Time Frame: 12 Week Time Point
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | 2.5% IL-1Ra | Placebo | 5% IL-1Ra
Number analyzed (Participants) | 30 | 30 | 15
Seconds | 4.5 (2.8) | 4.4 (2.3) | 3.9 (2.0)

3. Primary Outcome: Corneal Fluorescein Staining Score
Description: Is used to assess the level of corneal epitheliopathy that is related to dry eye disease. The CFS scale ranges from 0 to 15 scale, with 0 representing the minimum level of corneal epitheliopathy and 15 representing the maximum level of epitheliopathy.
Time Frame: 12 Week Time Point
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 2.5% IL-1Ra | Placebo | 5% IL-1Ra
Number analyzed (Participants) | 30 | 30 | 15
Units on a scale | 0.9 (0.7) | 1.4 (1.1) | 1.4 (0.8)

4. Primary Outcome: Ocular Surface Disease Index (OSDI)
Description: The Ocular Surface Disease Index (OSDI) is a 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning. The 12 items of the OSDI questionnaire are graded on a scale of 0 to 4, where 0 indicates none of the time; 1, some of the time; 2, half of the time; 3, most of the time; and 4, all of the time. The total OSDI score is then calculated on the basis of the following formula: OSDI=[(sum of scores for all questions answered) x 100]/[(total number of questions answered) x 4].
  Thus, the OSDI is scored on a scale of 0 to 100, with higher scores representing greater disability. A negative change from baseline indicated an improvement in vision-related functioning.
  OSDI was assessed on the Baseline Visit, Week 2, Week 6, Week 12, Week 16. Change indicated represents change from Baseline to Week 12.
Time Frame: Baseline and 12 Week Time Point data
Population: The OSDI analysis for this study is based on a standard intention-to-treat analysis with each study participant analyzed with respect to the randomized treatment assignment, regardless of eventual compliance.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Anakinra 2.5% Topical Ophthalmic Solution: In this study, the OSDI was assessed for patients taking Anakinra (KINERET) 2.5%. The outcome presented is a number that represents the percent change in OSDI score from baseline to week 12.
- Artificial Tear Topical Ophthalmic Solution: The OSDI was assessed for patients taking placebo. The outcome presented is a number that represents the percent change in OSDI score from baseline to week 12.
- Anakinra 5% Topical Ophthalmic Solution: The OSDI was assessed for patients taking Anakinra (KINERET) 5%. The outcome presented is a number that represents the percent change in OSDI score from baseline to week 12.
Arm/Group | Anakinra 2.5% Topical Ophthalmic Solution | Artificial Tear Topical Ophthalmic Solution | Anakinra 5% Topical Ophthalmic Solution
Number analyzed (Participants) | 30 | 30 | 15
units on a scale | 31.8 (24.1) | 41.8 (24.1) | 31.7 (19.0)

ADVERSE EVENTS:
Time Frame: 16 Weeks
Arm/Group | 2.5% IL-1Ra | Placebo | 5% IL-1Ra
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/30 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30 | 0/15
Other Adverse Events (participants affected / at risk) | 11/30 | 17/30 | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5% IL-1Ra (N=30) | Placebo (N=30) | 5% IL-1Ra (N=15)
Death (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Subject died due to complications resulting from chronic myelocytic leukemia
OTHER ADVERSE EVENTS (reported when occurring in more than 3.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5% IL-1Ra (N=30) | Placebo (N=30) | 5% IL-1Ra (N=15)
Stinging Eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Burning Eye (Eye disorders) | 1 (1) | 3 (3) | 0 (0)
Grittiness (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Itching Eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 2 (2) | 2 (2) | 1 (1)
Epiphora (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Discomfort (unspecific) (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eyelid Irritation (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Pingueculitis (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Episcleritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes